CLINICAL TRIAL: NCT05775172
Title: Gastric Myoelectric Activity, Inflammatory, Dietary, and Body Composition Changes During Weight Loss Via Bariatric Surgery and Lifestyle Modification
Brief Title: Weight Loss Via Bariatric Surgery and Lifestyle Modification
Status: Completed | Type: Observational
Sponsor: King Saud University (Other)
Collaborators: King AbdulAziz City for Science and Technology (Other)
Responsible Party: Principal Investigator, Mahmoud Abulmeaty, M.D., FACN., Professor, King Saud University
Other Study IDs: BSvsLS
Record Dates: First submitted 2023-03-03; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Obesity; Weight Loss
Keywords: gastric myoelectric activity; Inflammatory; bariatric surgery; lifestyle intervention; weight loss; body composition
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Waitlist control: Waitlist control (C group n=30) did not achieve any significant weight loss and did not follow lifestyle intervention
  Interventions: Other: Control
- Lifestyle intervention: Lifestyle intervention (LS group, n=22) follows multimodal lifestyle intervention in form of 500-100 kcal deficit , gradual physical activity and some behavioral modifications
  Interventions: Dietary Supplement: Lifestyle intervention
- Bariatric surgery: Bariatric surgery (BS group n=27) undergoes laparoscopic sleeve gastrectomy
  Interventions: Procedure: Sleeve gastrectomy

INTERVENTIONS:
Procedure: Sleeve gastrectomy — laparoscopic sleeve gastrectomy was done under general anesthesia by the same surgeon in the SBAHC. Routine preoperative, and postoperative care (including early post-operative dietary management) were done. Baseline assessment was taken within the last week before the surgery during the preoperative preparation and the final assessment was recorded 6 months after the surgery date.
  Groups: Bariatric surgery
Dietary Supplement: Lifestyle intervention — balanced 500 to 1000-calorie-deficit diet, personalized physical activity plan, and customized behavioral modification
  Groups: Lifestyle intervention
Other: Control — No interventions were applied
  Groups: Waitlist control

SUMMARY:
Gastric myoelectric, inflammatory, and hormonal responses, body compositional, energy expenditure, and metabolic changes during the development of obesity and the weight loss process are underinvestigated. This project studied the myoelectrical inflammatory and hormonal responses of the stomach, in addition to energy expenditure and body composition changes during weight loss via bariatric surgery and lifestyle intervention.

DETAILED DESCRIPTION:
Gastric myoelectric, inflammatory, and hormonal responses, body compositional, energy expenditure, and metabolic changes during the development of obesity and the weight loss process are underinvestigated. This project studied the myoelectrical, inflammatory, and hormonal responses of the stomach, in addition to energy expenditure and body composition changes during weight loss via bariatric surgery and lifestyle intervention.

Methods: We recruited 79 participants who were assigned to three groups: bariatric surgery (BS group n=27), lifestyle intervention (LS group, n=22), and waitlist control (C group n=30). For all participants, electrogastrography, inflammatory cytokines, gastric hormones analysis, body composition analysis, energy expenditure, and dietary assessment were done at baseline and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 35 kg/m2,
* Being free of any acute medical condition, inflammatory conditions, malignancy, or psychiatric disorders

Exclusion Criteria:

* Taking weight-losing pharmacotherapy
* Who underwent previous bariatric surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A total of 79 participants were randomly assigned to three groups: bariatric surgery (BS group n=27), lifestyle intervention (LS group, n=22), and waitlist control (C group n=30). The participants in the three groups were similar in BMI (>35 kg/m2), age (18-40 years), and gender. Inclusion criteria included BMI > 35 kg/m2, and being free of any acute medical condition, malignancy, or psychiatric disorders. Participants taking weight-losing pharmacotherapy or who underwent previous bariatric surgery were excluded. For all participants, electrogastrography, inflammatory cytokines measurements, body composition analysis, dietary assessment, and indirect calorimetry (as described in objective 1) were done at baseline, and after 6 months.
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
Gastric myoelectric activity | 6 months
  The gastric myoelectric activity was measured in fasting (for 10 mins) and post-prandial state (for 30 mins) using a multichannel electrogastrography (EGG) with a water load satiety test
Inflammatory changes | 6 months
  Serum levels of inflammatory markers involving interleukin-6 (IL-6), tumor necrosis factor-α (TNF-α), C-reactive protein (CRP), and monocyte chemoattractant protein (MCP-1),
Body composition measurement | 6 MONTHS
  Body composition was analyzed via a multi-Frequency segmental bioelectric impedance analysis monitor
Resting Energy Expenditure | 6 MONTHS
  Resting metabolic rate (RMR) was measured by the automated metabolic cart indirect calorimetry (IC) using a standard canopy hood
hormonal analysis | 6 Months
  serum levels of ghrelin, gastrin, and irisin (ELISA kits MyBiosource, San Diego, CA, USA; Catalog numbers: MBS2700428, MBS264399, MBS2600406, respectively).

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Abulmeaty, Principal Investigator — King Saud University
Locations (1):
- College of Applied Medical Sciences, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No